CLINICAL TRIAL: NCT01411657
Title: NT-501 CNTF Implant for Ischemic Optic Neuropathy: Safety, Neuroprotection and Neuroenhancement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey L Goldberg (Other)
Responsible Party: Sponsor-Investigator, Jeffrey L Goldberg, Associate Professor of Ophthalmology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090300
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Optic Neuropathy/Optic Nerve Stroke
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NT-501 CNTF Implant (Experimental): Patients will receive single NT-501 CNTF implant in one eye
  Interventions: Drug: NT-501 CNTF Implant

INTERVENTIONS:
Drug: NT-501 CNTF Implant — Single implantation of CNTF-secreting NT-501 device into one eye

SUMMARY:
Ciliary Neurotrophic Factor (CNTF) has been demonstrated in multiple preclinical models to enhance survival and regeneration of retinal ganglion cells, the retinal neurons injured in diseases like ischemic optic neuropathy/optic nerve stroke. We hypothesize that CNTF delivery to the human eye will provide neuroprotection (prevent loss of vision) and neuroenhancement (improve vision indices) in ischemic optic neuropathy. Patients in the trial will receive an NT-501 CNTF implant (made by Neurotech) into one eye, and will be carefully followed to evaluate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* age 40 years or older
* must understand and sign the informed consent
* must be medically able to undergo ophthalmic surgery for the NT-501 device insertion and possible removal, as well as the testing required.
* diagnosis of ischemic optic neuropathy characterized by (a) non-arteritic subtype, including a normal ESR and CRP; (b) syndrome of acute unilateral visual loss with documented optic nerve head edema but without significant pain; (c) a relative afferent papillary defect in the affected eye, and a decrease of best-corrected visual acuity to 20/40 or worse in the affected eye, and detectable loss on visual field testing consistent with nerve fiber visual field defect but retaining measurable residual visual field preservation.

Exclusion Criteria:

* other corneal, lens, optic nerve or retinal disease causing vision loss,
* blind in one eye
* requirement of acyclovir and/or related products during study
* receiving systemic steroids or other immunosuppressive medications.
* pregnant or lactating.
* considered immunodeficient or has a known history of human immunodeficiency virus (HIV)
* on chemotherapy, or a history of malignancy, UNLESS it was treated successfully 2 years prior to inclusion in the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety: Number of patients with adverse events | 18 months
  Safety will be evaluated by determining the number of patients with adverse events, including loss of vision, visual field, or retinal/optic nerve structure, and ocular complications such as pain and inflammation.

SECONDARY OUTCOMES:
Functional Efficacy: Vision, Visual Field, Pattern Electroretinogram, Visual Field Questionnaire-25 | 18 months
Structural efficacy: Nerve fiber layer, optic nerve topography | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bascom Palmer Eye Institute, University of Miami Miller School of Medicine, Miami, Florida, United States